CLINICAL TRIAL: NCT06148064
Title: EFFECT OF LOW-LEVEL LASER THERAPY ON STABILITY OF DENTAL IMPLANTS PLACED IN A FRESH EXTRACTED SOCKET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #2/3/2023
Record Dates: First submitted 2023-11-17; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Dental Implant Stability

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaplug application with low level laser application. (Experimental)
  Interventions: Other: Collaplug with low level laser
- Collaplug application (Active Comparator)
  Interventions: Other: Collaplug

INTERVENTIONS:
Other: Collaplug with low level laser — Immediate implant placement with applying a collaplug material in the jumping gap followed by low level laser application using Siro laser (660 nm, avg. power density: 0.5-WATT) circular spot diameter and area: 0.71 cm/0.4cm2) applied in six points in contact mode with peri-implant soft tissue (1.23 minutes in each point of application; dose per point 11 J) before bone perforation and after suturing.
  Arms: Collaplug application with low level laser application.
Other: Collaplug — Implant of suitable diameter and height was placed in the fresh extracted socket immediately after extraction and the jumping gap was augmented by the collaplug followed by healing abutment placement.
  Arms: Collaplug application

SUMMARY:
Aim of the study was to evaluate the effect of low-level laser therapy (LLLT) (660nm laser diode 0.5W) on implant stability and crestal bone loss in implants inserted in freshly extracted sockets augmented by Collaplug in the jumping gap.

ELIGIBILITY:
Inclusion Criteria:

* 1. Any non-restorable hopeless tooth: badly decayed tooth that cannot be restored. Tooth with failed endodontic treatment and tooth with longitudinal fracture.
* Type I post-extraction sockets with all bony walls intact.
* No signs of active periodontal disease in the selected tooth.

Exclusion Criteria:

* The presence of any systemic disease that could complicate bone or soft tissue healing after immediate implant placement.
* The presence of acute periapical infection.
* The presence of any local factor that may interfere with extraction as tooth ankyloses.
* Subjects who had undergone therapeutical radiation.
* Patients who had been subjected to or who were under bisphosphonate therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Implant stability | up to 3 months
  Implant stability was measured by OSSTELL at 4 different levels (buccal, lingual, mesial, and distal). Implant Stability Quotient, is a scale from 1 to 100 and is a measure of the stability of an implant. Higher levels indicate greater stability.
Crestal bone loss | up to 3 months
  Crestal bone loss was assessed using cone beam computed tomography (CBCT) by measuring the distance from the bone crest to the implant apex from mesial, distal, lingual and buccal aspects intraoperatively. Crestal bone loss up to 1.5 mm is considered a normal early finding through the first year after implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Nermine A Elnakib, BDS, Principal Investigator — Alexandria University; Maha R Talaab, PhD, Study Chair — Alexandria University; Nayrouz A Metwally, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt